CLINICAL TRIAL: NCT05772507
Title: Assessment of the Efficacy and Tolerance of URGO AWC_008 and URGO AWC_022 Dressings in Local Management of Acute and Chronic Wounds at Risk of Local Infection or With Clinical Signs of Local Infection
Brief Title: Efficacy and Tolerance of URGO AWC_008 and URGO AWC_022 Dressings (EXPANSION)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDRCB no.: 2022-A00862-41
Record Dates: First submitted 2023-03-02; First posted 2023-03-16 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer; Pressure Ulcer; Wound Infection; Acute Wounds
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer; Wound Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- medical device under investigation (Experimental): URGO AWC_008 or URGO AWC_022 dressing. These 2 dressings are similar and only the adhesive constitutes a difference. The choice of study dressing will be left to the discretion of the investigator during the treatment of the patient, depending on the nature of the wound and the condition of the peri-wound skin.
  Interventions: Device: URGO AWC_008 dressing or URGO AWC_022 dressing

INTERVENTIONS:
Device: URGO AWC_008 dressing or URGO AWC_022 dressing — local management of acute or chronic wounds

SUMMARY:
Evaluation of the efficacy (wound epithelialization and time to closure) and tolerance (emergence and nature of adverse event) of the new URGO AWC_008 and URGO AWC_022 dressings in local management of acute and chronic wounds at risk of local infection or with clinical signs of local infection

DETAILED DESCRIPTION:
prospective multicenter, non comparative clinical investigation

This is a prospective multicenter, non comparative open-label, clinical investigation conducted in patients with acute and chronic wounds at risk of local infection or with clinical signs of local infection.

This study is carried out in France and Spain in around 30 investigator sites. A total of 85 patients meeting the eligibility criteria will be included. The patients will be followed for 4 weeks and a total of 5 clinical evaluations will be carried out by the investigating centers.

A planimetric survey of the studied wounds is carried out during the initial assessment of the wound (Day 0) and at each assessment provided for in the protocol (Week 1, Week 2, Week 3 and Week 4).

ELIGIBILITY:
Inclusion Criteria :

Related to all wounds :

* Adult patient having given free, informed and written consent
* Patient affiliated to a social security insurance scheme (applicable For France),
* Inpatient or outpatient who can be followed by the same investigative team throughout the investigation,
* Acute wound (burn, traumatic wound, unstitched surgical wound) or chronic wound (leg ulcer, pressure ulcer, diabetic foot ulcer),
* Wound whose surface can be covered by a single dressing,
* Wound at least 3 cm from any edge of another wound.

Related to acute wounds, leg ulcer, pressure ulcer:

Patient whose studied wound presents a risk of local infection (based on modified W.A.R. score ≥ 3 points) or with at least 3 of the following clinical signs:

* Pain (spontaneous, pressure pain or increased pain),
* Peri-wound erythema,
* Oedema, induration or swelling,
* Odour (increase, change),
* Exudate (colour modification or increase of exudate),
* Local warmth,
* Hypergranulation,
* Bleeding, friable granulation tissue,
* Stagnant healing/wound deterioration.

Related to diabetic foot ulcer :

Patient whose studied wound presents a risk of local infection (based on modified W.A.R. score ≥ 3 points) or with at least 2 of the following clinical signs:

* Pain (spontaneous, pressure pain or increased pain),
* Peri-wound erythema between 0.5-2.0 cm around the wound,
* Oedema, induration or swelling,
* Odour (increase, change),
* Exudate (colour modification or increase of exudate),
* Local warmth,
* Hypergranulation,
* Bleeding, friable granulation tissue,
* Stagnant healing/wound deterioration,

Exclusion Criteria:

* Patient with a wound for which treatment in a hyperbaric chamber is planned within 4 weeks following inclusion,
* Patient with a serious general condition, that could lead to withdrawal from the trial before four weeks of treatment,
* Patient who has experienced an acute ischaemic event (acute myocardial infarction or stroke) during the 3 months prior to inclusion in the investigation,
* Patient with a systemic infection
* Wound totally or partially covered on its surface with a black plaque of necrosis,
* Cancerous wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
relative wound area reduction (RWAR) | 4 week treatment period
  changes in the area of wounds after 4 weeks of treatment.

SECONDARY OUTCOMES:
percentage of patients whose wound has healed | 4 week treatment period
  Complete closure of the Venous Leg Ulcer (VLU) - Healing of the wound is defined by 100% re-epithelialization of the wound
Nature and incidence of Treatment Adverse Effects as assessed in percentage for each dressing | 4 week treatment period
  Safety analysis with nature and number of adverse event related to the use of the dressings (serious/ non-serious)

CONTACTS AND LOCATIONS:
Locations (1):
- URGO, Dijon, France

IPD SHARING:
Plan to Share IPD: No